CLINICAL TRIAL: NCT03973723
Title: Long-term Results of Plasma Epstein-Barr Virus DNA Monitoring In Nasopharyngeal Carcinoma After Curative Treatment
Brief Title: Plasma EBV DNA Monitoring in Post-treatment NPC Patients
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CG11133
Record Dates: First submitted 2019-06-03; First posted 2019-06-04 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Nasopharyngeal Carcinoma; NPC; EBV; Radiotherapy
Keywords: Nasopharyngeal Carcinoma; NPC; EBV; Radiotherapy; Plasma Epstein-Barr virus DNA
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and check plasma EBV DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with NPC after treatment: All patients with NPC without distant metastases who receiving adequate RT dose

SUMMARY:
Continuous regular monitoring of plasma EBV DNA in nasopharyngeal carcinoma (NPC) after treatment have rarely been investigated. The investigators try to analyze the long-term observational results (role in early relapse detection and impact on survival) in NPC patients after curative treatment.

DETAILED DESCRIPTION:
The investigators enrolled 441 NPC patients who had finished finished curative radiotherapy with/without chemotherapy and no recurrence/metastasis before entry this study from five hospitals in Taiwan. Blood samples were collected on the day of enrollment and monitored once every 2-3 months for plasma EBV DNA measurement. After long-term observation, we analyze the impact of continuous plasma EBV DNA monitoring on the early dection of tumor relapse and do risk grouping for survival analyses according to the blood test results.

ELIGIBILITY:
Inclusion criteria

* histologically-proven nasopharyngeal carcinoma without distant metastasis (M0) at initial presentation
* finished curative radiotherapy (with/without chemotherapy) within 3 years

Exclusion criteria

* no occurrence of documented recurrence/metastasis before entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with NPC who were treated at 5 hospitals (Taichung Veterans General Hospital, Taichung; Yuan's General Hospital, Kaohsiung; National Cheng Kung University Hospital, Tainan; Kaohsiung Medical University Hospital, Kaohsiung; Taipei Medical University Hospital, Taipei; Taiwan)
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Time interval from the date of abnormal blood test to the date of clinically documented tumor relapse | Five years
  From the end of treatment to any time when abnormal blood test is fund

SECONDARY OUTCOMES:
Overall survival (OS) | Five years
  Overall survival was calculated from the day of enrollment until death or the last follow-up visit
Event-free survival (EFS) | Five years
  Event-free survival was calculated from the day of enrollment until the date of first occurrence of tumor relapse (local, regional, or distant failures) or the last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ching Lin, M.D.,PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee AW, Poon YF, Foo W, Law SC, Cheung FK, Chan DK, Tung SY, Thaw M, Ho JH. Retrospective analysis of 5037 patients with nasopharyngeal carcinoma treated during 1976-1985: overall survival and patterns of failure. Int J Radiat Oncol Biol Phys. 1992;23(2):261-70. doi: 10.1016/0360-3016(92)90740-9. PMID 1587745
- [Background] Jiong L, Berrino F, Coebergh JW. Variation in survival for adults with nasopharyngeal cancer in Europe, 1978-1989. EUROCARE Working Group. Eur J Cancer. 1998 Dec;34(14 Spec No):2162-6. doi: 10.1016/s0959-8049(98)00322-0. PMID 10070282
- [Background] Lin JC, Jan JS, Hsu CY, Jiang RS, Wang WY. Outpatient weekly neoadjuvant chemotherapy followed by radiotherapy for advanced nasopharyngeal carcinoma: high complete response and low toxicity rates. Br J Cancer. 2003 Jan 27;88(2):187-94. doi: 10.1038/sj.bjc.6600716. PMID 12610501
- [Background] Lin JC, Jan JS, Hsu CY, Liang WM, Jiang RS, Wang WY. Phase III study of concurrent chemoradiotherapy versus radiotherapy alone for advanced nasopharyngeal carcinoma: positive effect on overall and progression-free survival. J Clin Oncol. 2003 Feb 15;21(4):631-7. doi: 10.1200/JCO.2003.06.158. PMID 12586799
- [Background] Lin JC, Jan JS, Chen KY, Hsu CY, Liang WM, Wang WY. Outpatient weekly 24-hour infusional adjuvant chemotherapy of cisplatin, 5-fluorouracil, and leucovorin for high-risk nasopharyngeal carcinoma. Head Neck. 2003 Jun;25(6):438-50. doi: 10.1002/hed.10238. PMID 12784235
- [Background] Chan AT, Teo PM, Leung TW, Leung SF, Lee WY, Yeo W, Choi PH, Johnson PJ. A prospective randomized study of chemotherapy adjunctive to definitive radiotherapy in advanced nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 1995 Oct 15;33(3):569-77. doi: 10.1016/0360-3016(95)00218-N. PMID 7558945
- [Background] Cheng SH, Jian JJ, Tsai SY, Chan KY, Yen LK, Chu NM, Tan TD, Tsou MH, Huang AT. Prognostic features and treatment outcome in locoregionally advanced nasopharyngeal carcinoma following concurrent chemotherapy and radiotherapy. Int J Radiat Oncol Biol Phys. 1998 Jul 1;41(4):755-62. doi: 10.1016/s0360-3016(98)00092-3. PMID 9652835
- [Background] International Nasopharynx Cancer Study Group; VUMCA I Trial. Preliminary results of a randomized trial comparing neoadjuvant chemotherapy (cisplatin, epirubicin, bleomycin) plus radiotherapy vs. radiotherapy alone in stage IV(> or = N2, M0) undifferentiated nasopharyngeal carcinoma: a positive effect on progression-free survival. Int J Radiat Oncol Biol Phys. 1996 Jun 1;35(3):463-9. doi: 10.1016/s0360-3016(96)80007-1. PMID 8655368